CLINICAL TRIAL: NCT05578742
Title: Effect of PEEP on Ventilartion/Perfusion Ratios According to Different Phenotypes in Patients With ARDS (France)
Brief Title: V/Q Matching Variations With PEEP in ARDS According to Compliance-based Phenotypes (France)
Acronym: MISMATCHED FR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-A00649-34
Record Dates: First submitted 2022-09-27; First posted 2022-10-13 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: ARDS
Keywords: pulmonary perfusion; ventilation-perfusion mismatch; compliance; recruitability
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Intervention Model Description: Fifty patients will be enrolled, divided into 2 groups (n=26 each) according to a dynamic balanced sampling based on normalized respiratory system elastance (ERS) measured at PEEP 5 cmH2O with Vt 6-7 ml/kg PBW (<2 cmH2O.mL-1.kg-1 vs. ≥2 cmH2O.mL-1.kg-1). Enrolment into each study group will be closed at 26 patients.
  Then, patients will be randomized and allocated to one of the following strategies:
  * Strategy A: PEEP 15 cmH2O → PEEP 5 cmH2O
  * Strategy B: PEEP 5 cmH2O → PEEP 15 cmH2O
  A parallel study will be conducted in Italy, to reach 50 more patients. Data will be shared between these two studies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strategy A: PEEP 15 cmH2O → PEEP 5 cmH2O (Experimental)
  Interventions: Procedure: PEEP decrease
- Strategy B: PEEP 5 cmH2O → PEEP 15 cmH2O (Active Comparator)
  Interventions: Procedure: PEEP increase

INTERVENTIONS:
Procedure: PEEP increase — Positive End Expiratory Pressure (PEEP) will be increased from 5 to 15 cmH2O.
  Arms: Strategy B: PEEP 5 cmH2O → PEEP 15 cmH2O
Procedure: PEEP decrease — Positive End Expiratory Pressure (PEEP) will be decreased from 15 to 5 cmH2O.
  Arms: Strategy A: PEEP 15 cmH2O → PEEP 5 cmH2O

SUMMARY:
This study aim to compare the effect of Positive End Expiratory Pressure (PEEP) on ventilation/perfusion mismatch in two phenotypes of patients with moderate-to-severe Acute Respiratory Distress Syndrome (ARDS), characterized by their respiratory system elastance (Ers). Ventilation/perfusion mismatch will be assessed by Electrical Impedance Tomography (EIT).

DETAILED DESCRIPTION:
Acute Respiratory Distress Syndrome (ARDS) is characterized by hypoxemia caused by inflammatory lung injury. Recent studies showed an important variability in ARDS phenotypes . The recent COVID-19 crisis highlighted the presence of ARDS patients with severe hypoxemia and normal respiratory system compliance, and retrospective series confirmed the existence of this atypical ARDS pattern also in non-COVID etiologies.

The dissociation between mechanics and hypoxemia may be related to a specific diversity in the pattern of ventilation-perfusion matching (V/Q matching) among patients with normal compliance and ARDS. In patients with low compliance, V/Q mismatch may be characterized by right-to-left shunt, secondary to collapse of the gravity-dependent regions; while, in patients with normal compliance, V/Q mismatch may show a redistribution of blood flow to hypo-ventilated lung areas by larger dead space and impaired hypoxic vasoconstriction.

These differences may also influence the response to PEEP in terms of gas exchange and lung protection . It may also explain the failure for high PEEP levels to improve significantly mortality in the global ARDS population (i.e., with patients' selection only based on hypoxemia).

Electrical Impedance Tomography (EIT) is a device allowing to assess ventilation and perfusion distribution. Thus, EIT can be used to evaluate global and regional V/Q matching, and could be used to understand mechanisms of hypoxemia, especially in patients with normal mechanics and ARDS.

The aim of this study is to assess V/Q matching according to these different ARDS phenotypes, and to evaluate the effects of PEEP in each one.

ELIGIBILITY:
Inclusion criteria:

* intubated patients with moderate and severe ARDS (Berlin definition, PaO2/FiO2 ≤200 mmHg at PEEP 5 cmH2O)
* undergoing deep sedation
* on controlled mechanical ventilation
* between 24 hours and 5 days after intubation.

Exclusion criteria:

* age <18 years old; pregnancy
* patient undergoing legal protection
* contra-indications to EIT (e. g. severe chest trauma or wounds)
* pneumothorax; patient undergoing ECMO
* patient with BMI ≥35 kg/m2
* hemodynamic instability with MAP <60 mmHg despite vasopressors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Difference in ventilation/perfusion mismatch between PEEP 5 and 15 cmH2O according to the two studied phenotypes | immediately after each intervention
  Ventilation/perfusion (V/Q) mismatch will be assessed by Electrical Impedance Tomography (EIT). Mismatch is expressed in %. Comparison between phenotype with higher and lower elastance will be performed.

SECONDARY OUTCOMES:
Difference in respiratory mechanics between PEEP 5 and 15 cmH2O according to the two studied phenotypes | immediately after each intervention
  Plateau pressure and total PEEP will be aggregated to compute driving pressure (Plateau pressure minus total PEEP, all in cmH2O). Respiratory system compliance will be computed by dividing tidal volume by driving pressure (in mL.cmH2O-1; respiratory system resistance will be computed as the inverse of compliance; all these values will be assessed and compared between the two PEEP levels. Comparison between phenotype with higher and lower elastance will be performed.
Difference in oxygenation between PEEP 5 and 15 cmH2O according to the two studied phenotypes | immediately after each intervention
  PaO2 (in mmHg) will be assessed and compared between the two PEEP levels. Comparison between phenotype with higher and lower elastance will be performed.
Difference in carbon clearance between PEEP 5 and 15 cmH2O according to the two studied phenotypes | immediately after each intervention
  PaCO2 (in mmHg) will be assessed and compared between the two PEEP levels. Ventilatory ratio (no unit) will be derived from the PaCO2 values. Comparison between phenotype with higher and lower elastance will be performed.
Difference in dead space measured by capnometric volumetry between PEEP 5 and 15 cmH2O according to the two studied phenotypes | immediately after each intervention
  VCO2 (measured by Vcap, in mmHg) will be assessed and compared between the two PEEP levels. Comparison between phenotype with higher and lower elastance will be performed.
Difference in dead space measured by calorimetry between PEEP 5 and 15 cmH2O according to the two studied phenotypes | immediately after each intervention
  VCO2 (measured by calorimetry, in mmHg) will be assessed and compared between the two PEEP levels. Comparison between phenotype with higher and lower elastance will be performed.
Difference in venous oxygen saturation between PEEP 5 and 15 cmH2O according to the two studied phenotypes | immediately after each intervention
  SvO2 (in %) will be assessed and compared between the two PEEP levels. Comparison between phenotype with higher and lower elastance will be performed.
Correlation between V/Q mismatch markers and recruitability | immediately after each intervention
  Recruitability will be assessed between 15 and 5 cmH2O by respiratory mechanics and EIT, as the recruited volumes value (in mL). R/I ratio will be derived from these data (no unit). V/Q mismatch will be computed by EIT, and expressed in %. Correlation will be performed by linear regression.
Correlations between V/Q mismatch assessed by EIT and dead space markers | immediately after each intervention
  Dead space will be assessed by volumetric capnography (if available), venrtilatory ratio, and calorimetriy (if available). V/Q mismatch will be computed by EIT, and expressed in %. Correlation will be performed by linear regression.
Correlations between V.Q mismacth and overdisension and lung collapsus | immediately after each intervention
  Overdistension (%) and lung collapsus (%) will be assessed during the Step 3, by EIT. These two values cannot be measured separately. V/Q mismatch will be computed by EIT, and expressed in %. Correlation will be performed by linear regression.
Difference in stress index between PEEP 5 and 15 cmH2O according to the two studied phenotypes | immediately after each intervention
  stress index (no unit) will be assessed and compared between the two PEEP levels. Comparison between phenotype with higher and lower elastance will be performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Angers Hospital, Angers, Maine et Loire, France

IPD SHARING:
Plan to Share IPD: Yes